CLINICAL TRIAL: NCT00341029
Title: Measurement of Cytogenetic Endpoints in Lymphocytes of Children Diagnosed With Attention Deficit/Hyperactivity Disorder (ADHD) and Treated With Methylphenidate or Adderall
Brief Title: Genetic Measurements in Blood Cells of Children Taking Adderall or Methylphenidate
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906045; 06-E-N045
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-26

CONDITIONS: Attention Deficit Hyperactivity Disorder; ADHD
Keywords: Longitudinal Study; Chromosomal Effects; Sister Chromatid Exchanges; Micronuclei; Stimulants; Attention Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

SUMMARY:
This study, conducted at Duke University in Durham, NC, will determine whether the drugs Adderall and methylphenidate affect the genetic material of children with attention deficit hyperactivity disorder (ADHD). One small study has shown that taking methylphenidate for ADHD may result in higher levels of certain types of changes to the genetic material contained in white blood cells. The changes seen are not directly linked to increased risk of disease, but indicate a possibility that other kinds of damage that may be linked to increased disease may result from taking methylphenidate. The study will also examine whether these types of changes might occur in children treated with Adderall .

Children between the ages of 6 and 12 with symptoms of ADHD may be eligible for this study. Candidates are screened with a medical history, psychiatric examination, IQ test, physical examination, and electrocardiogram. Parents and teachers complete questionnaires to rate the severity of the child's ADHD. Qualified children who are diagnosed with ADHD and who are appropriate candidates for treatment with either Adderall or methylphenidate-based drugs (e.g., Concerta, Metadate, Focalin, Ritalin or Ritalin LA) may be selected for this study.

At a baseline visit (Visit 0), parents complete questionnaires that rate the severity of their child's ADHD. The children have their vital signs checked (pulse, blood pressure, breathing rate, height, weight and temperature) and have a blood sample drawn. The children are then randomly assigned to treatment with either Adderall or a methylphenidate product. After the baseline visit, participants undergo the following tests and procedures:

Dose Optimization Visits (visits 1-4)

In the first 4 weeks of the study, the dose of methylphenidate or Adderall is adjusted weekly until doctors determine the dose strength that works best for the individual child. In addition, the following procedures are done at each visit:

* Child's vital signs are checked.
* Parents complete a questionnaire about the severity of the child's ADHD.
* Parent and child describe the impact of symptoms on the child's functioning.
* Parents complete forms about common side effects of the study drug.

Follow-up Visits (visits 5-6)

Children return to the clinic once a month to assess their health and further adjust their medication dose, if needed. The visits are similar to those during the dose optimization period, with the following additional procedures at visit 6:

* A blood sample is obtained to measure whether the medication has affected the child's genetic material.
* A physical examination is done to check child's health.
* Information is provided parents to assist in planning for child's treatment after the study.

DETAILED DESCRIPTION:
Design: Longitudinal observational study of pediatric ADHD patients, any subtype. This study is part of a large comprehensive investigation initiated and funded by the National Institute of Child Health and Human Development to aid in the understanding of a reported association of methylphenidate treatment and elevated frequencies of some types of chromosome damage.

Population: 60 diagnosed ADHD children, age range 6-12 years inclusive, for whom pharmacological treatment with stimulant medication is indicated. 30 children will initiate treatment with a methylphenidate-based product and 30 will initiate treatment with Adderall or Adderall-XR. Study group assignment will be randomized, as these two drugs are considered by the clinical community to be fully interchangeable.

Primary Objective: To determine the frequency of micronuclei (markers of numerical or structural chromosomal damage), sister chromatid exchanges (indicators of DNA damage), and chromosomal aberrations in lymphocytes of pediatric ADHD patients prior to and after 3 months of uninterrupted drug therapy. These endpoints, and the time frame, are compatible with investigating effects during the initiation phase of treatment; additional studies by other NIH institutes (NIMH, CDC) will investigate effects after chronic treatment with stimulant medications so that a comprehensive picture of the potential for treatment-induced chromosomal damage in ADHD subjects is obtained.

Secondary Objective: In pediatric ADHD patients treated with a methylphenidate-based product or Adderall, to determine if flow cytometric measurement of the frequency of micronucleated erythrocytes can serve as a biomarker of cytogenetic damage in lymphocytes evaluated by standard light microscope techniques.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children of either sex, and of any ethnicity and economic status, age 6-12 years inclusive, who are diagnosed with ADHD, who are drug na ve, and who are determined by the study psychiatrist to be appropriate candidates for pharmacological therapy with either Adderall or methylphenidate-based drugs.

Child must be in good health as determined by medical history, physical examination and electrocardiogram (ECG).

EXCLUSION CRITERIA:

Children less than 6 years of age.

Children more than 12 years of age.

Children not determined to meet the comprehensive criteria for diagnosis of ADHD.

Children with co-morbid psychological conditions that would containdicate treatment with stimulant drugs.

Children who have previously undergone drug treatment for ADHD.

Children who have received diagnostic x-rays (not dental x-rays) within the past 3 months.

Female children who have had their first menstrual period.

Subjects who are not competent to provide consents.

Children determined by the study physician to be poor candidates for pharmacological therapy with Adderall or methylphenidate-based drugs.

Children with clinically significant abnormal electrocardiogram (ECG).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84
Dates: Start 2005-12-07; Primary Completion 2007-09-30 (Actual); Study Completion 2007-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Bonassi S, Hagmar L, Stromberg U, Montagud AH, Tinnerberg H, Forni A, Heikkila P, Wanders S, Wilhardt P, Hansteen IL, Knudsen LE, Norppa H. Chromosomal aberrations in lymphocytes predict human cancer independently of exposure to carcinogens. European Study Group on Cytogenetic Biomarkers and Health. Cancer Res. 2000 Mar 15;60(6):1619-25. PMID 10749131
- [Background] Bonassi S, Ugolini D, Kirsch-Volders M, Stromberg U, Vermeulen R, Tucker JD. Human population studies with cytogenetic biomarkers: review of the literature and future prospectives. Environ Mol Mutagen. 2005 Mar-Apr;45(2-3):258-70. doi: 10.1002/em.20115. PMID 15688363
- [Background] Dertinger SD, Torous DK, Hall NE, Murante FG, Gleason SE, Miller RK, Tometsko CR. Enumeration of micronucleated CD71-positive human reticulocytes with a single-laser flow cytometer. Mutat Res. 2002 Mar 25;515(1-2):3-14. doi: 10.1016/s1383-5718(02)00009-8. PMID 11909751
- [Derived] Witt KL, Shelby MD, Itchon-Ramos N, Faircloth M, Kissling GE, Chrisman AK, Ravi H, Murli H, Mattison DR, Kollins SH. Methylphenidate and amphetamine do not induce cytogenetic damage in lymphocytes of children with ADHD. J Am Acad Child Adolesc Psychiatry. 2008 Dec;47(12):1375-83. doi: 10.1097/CHI.0b013e3181893620. PMID 18978633